CLINICAL TRIAL: NCT06270134
Title: Dial-Bicarb Trial: Effects of a Lower vs. Higher Concentration of Dialysate Bicarbonate for People Receiving Maintenance Hemodialysis
Brief Title: Dial-Bicarb Trial: Effects of a Lower vs. Higher Concentration of Dialysate Bicarbonate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); ACT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14410
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Renal Failure; Hemodialysis
Keywords: bicarbonate; renal failure; kidney; pragmatic trial; maintenance hemodialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — Bicarbonates

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, two-arm, parallel-group, open-label, individual-randomized, superiority trial that will be conducted in hemodialysis units across Ontario. Patients at each dialysis unit will be randomly allocated into one of two study arms in a 1:1 ratio to receive a dialysate bicarbonate concentration of either 32 or 38 mmol/L.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower dialysate bicarbonate concentration (32 versus mmol/L) (Active Comparator): Patients at each dialysis unit will be randomly allocated into one of two study arms in a 1:1 ratio to receive a dialysate bicarbonate concentration of 32 mmol/L.
  Interventions: Other: Bicarbonate
- Higher dialysate bicarbonate concentration (38 mmol/L) (Active Comparator): Patients at each dialysis unit will be randomly allocated into one of two study arms in a 1:1 ratio to receive a dialysate bicarbonate concentration of 38 mmol/L.
  Interventions: Other: Bicarbonate

INTERVENTIONS:
Other: Bicarbonate — Bicarbonate is added to hemodialysis fluids to correct the metabolic acidosis that arises from kidney failure. Some dialysis units in Canada add bicarbonate to a level of 32 mmol/L, while other units add bicarbonate to a level of 38 mmol/L. It is unknown whether one level is better for people's health.

SUMMARY:
This is a pragmatic, two-arm, parallel-group, open-label, individual-randomized, superiority trial that will be conducted in hemodialysis units across Ontario. Patients at each dialysis unit will be randomly allocated into one of two study arms in a 1:1 ratio to receive a dialysate bicarbonate concentration of either 32 or 38 mmol/L. The intervention will be embedded into routine care and delivered by hemodialysis unit personnel.

DETAILED DESCRIPTION:
Background: Bicarbonate is added to hemodialysis fluids to correct the metabolic acidosis that arises from kidney failure. Some dialysis centres in Canada add bicarbonate to a level of 32 mmol/L, while other centres add bicarbonate to a level of 38 mmol/L. It is unknown whether one level is better for people's health.

Objective: In patients receiving maintenance hemodialysis, to determine if providing a lower versus higher concentration of dialysate bicarbonate (32 versus 38 mmol/L) alters the risk of outcomes important to patients and their care providers.

Design, Setting, and Participants: This is a pragmatic, two-arm, parallel-group, open-label, individual-randomized, superiority trial that will be conducted in hemodialysis centres across Ontario. Patients at each dialysis centre will be randomly allocated into one of two study arms in a 1:1 ratio to receive a dialysate bicarbonate concentration of either 32 or 38 mmol/L. The intervention will be embedded into routine care and delivered by hemodialysis centre personnel. The concentration of dialysate bicarbonate is altered for a hemodialysis session through a simple setting on the machine.

Altered approach to patient consent: The study team, which includes patient partners, proposes an opt-out altered approach to patient consent to receive the trial-assigned concentration of dialysate bicarbonate. This is under a framework that Dial-Bicarb fits the required parameters to do so, as constructed in Canada's Tri-Council Policy Statement-2 (TCPS-2) Article 3.7A.

Primary Outcome: Two primary outcomes, all-cause mortality and recurrent all-cause non-elective hospitalizations.

Secondary Outcomes: Cardiovascular-related hospitalizations, infection-related hospitalizations, and fractures.

Data Collection: This trial will obtain information on patient characteristics and outcomes from provincial healthcare administrative databases, which are already collected as part of routine healthcare.

Planned Analysis: Treatment effects will be reported as hazard ratios accounting for the number of events and total follow-up time within arms.

Potential Impact: If a lower concentration of dialysate bicarbonate is shown to be superior, it could be easily adopted as the standard of care by hemodialysis centres globally at little added cost. This change in practice could help reduce premature deaths and hospitalizations among the more than 2 million people on hemodialysis worldwide.

ELIGIBILITY:
Inclusion Criteria:

* The dialysis centre director and all nephrologists who provide care in the centre agree to trial participation.
* Adult patients 18 years of age and older, with a health card number, enter the trial after they receive hemodialysis for at least 90 days (about 3 months) so that patients with acute kidney injury who recover kidney function are excluded.

Exclusion Criteria:

- Participating centres are instructed that patients on in-centre nocturnal hemodialysis or in-centre frequent (greater than four times weekly) hemodialysis are not in the trial (and do not receive the allocated intervention), since these patients usually receive dialysate bicarbonate concentrations ≤32mmol/L as standard care (based on Ontario registry data, these modalities represent <5% of the hemodialysis patient population).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Non-elective hospitalizations | Duration of the study, 4 years.
  All-cause recurrent non-elective hospitalizations
Mortality | Duration of the study, 4 years.
  All-cause mortality

SECONDARY OUTCOMES:
Hospitalizations and fractures | Duration of the study, 4 years.
  Cardiovascular-related hospitalizations, infection-related hospitalizations, and fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, MD, Principal Investigator — LHSC

IPD SHARING:
Plan to Share IPD: No